CLINICAL TRIAL: NCT05186662
Title: Comparing the Efficacy of WeChat-based Patient Education and Conventional Patient Education in the Management of Helicobacter Pylori Eradication
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Professor, Director of gastroenterology department of Qilu hospital, Shandong University
Other Study IDs: 2021SDU-QILU-111
Record Dates: First submitted 2021-12-25; First posted 2022-01-11 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Helicobacter Pylori Infection Helicobacter Pylori Eradication Patient Education
Keywords: helicobacter pylori eradication patient education Wechat group
MeSH Terms: interventions — Patient Education as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- WeChat group
  Interventions: Other: patient education
- Control group
  Interventions: Other: patient education

INTERVENTIONS:
Other: patient education — patients in experimental group were asked to join a WeChat group, which was governed by experienced gastroenterologists. Relevant knowledge of H. pylori eradication was released in the group chat irregularly. Patients in WeChat group were allowed to ask questions at any time during the whole treatment process, soon afterwards, suggestions were given.
  Groups: WeChat group
Other: patient education — Patients in the control group received verbal education and a specifically designed printout with detailed instructions.
  Groups: Control group

SUMMARY:
we conducted a retrospective study to compare the efficacy of WeChat-based patient education and conventional patient education in the management of Helicobacter pylori eradication.

DETAILED DESCRIPTION:
This is a single-institute retrospective study comparing the efficacy of WeChat-based patient education and conventional patient education in the management of Helicobacter pylori eradication. We identified all patients aged between 18-75 years old and had been prescribed a 14-day course of bismuth-contained quadruple therapy for H. pylori infection in our outpatient clinics between 1 July 2019 and 31 July 2021. H. pylori infection was confirmed by any two positive outcomes of rapid urease test,13C-urea breath test (UBT) and histopathology. Patients who had H. pylori therapy history, using other therapeutic regimens or unwilling to take prescribed medications were excluded. Demographic data, treatment regimens, outcomes of therapy, adherence to therapy and adverse event were retrieved. The main indicator is eradication rate, as the secondary indicators are compliance and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18 and 75 years old and have not been treated before.

Exclusion Criteria:

* Patients who had H. pylori therapy history, using other therapeutic regimens or unwilling to take prescribed medications were excluded. Demographic data, treatment regimens, outcomes of therapy, adherence to therapy and adverse event were retrieved.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients aged between 18-75 years old and had been prescribed a 14-day course of bismuth-contained quadruple therapy for H. pylori infection in our outpatient clinics between 1 July 2019 and 31 July 2021. H. pylori infection was confirmed by any two positive outcomes of rapid urease test,13C-urea breath test (UBT) and histopathology. Patients who had H. pylori therapy history, using other therapeutic regimens or unwilling to take prescribed medications were excluded.
Sampling Method: Probability Sample
Enrollment: 1017 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
eradication rate | 2 months
  Six weeks after completion of treatment，numbers of patients get H.pylori eradicated supported by negative 13C-UBT results will be investigated by an independent researcher.Then eradication rate in each group will be calculated by using intention-to-treat analysis and per-protocol analysis.

SECONDARY OUTCOMES:
compliance | 14 days
  compliance was evaluated by assessing the total pills patients have taken.Compliance was defined as good when more than 80% or less than 120% of the total pills were taken.
prevalence of adverse events | 14 days
  At the follow-up, adverse events complained by patients will be recorded by an independent researcher，meanwhile a 8 point visual analog scale (VAS) was used to evaluate severity of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hosipital, Jinan, Shandong, China